CLINICAL TRIAL: NCT03433989
Title: Impact of Post-Traumatic Stress Disorder After Pregnancy Loss After 12 Weeks of Gestation (Termination of Pregnancy , Stillbirth, Late Miscarriage)
Brief Title: ACTRAMAT-D: Impact of Post-Traumatic Stress Disorder After Pregnancy Loss After 12 Weeks of Gestation
Acronym: ACTRAMAT-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A02588-45
Record Dates: First submitted 2018-01-12; First posted 2018-02-15 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2019-12

CONDITIONS: Pregnancy Loss
Keywords: Post-Traumatic Stress Disorder; Pregnancy loss
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, epidemiological, descriptive and analytical study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnosis and follow up arm (Experimental)
  Interventions: Diagnostic Test: telephone interview

INTERVENTIONS:
Diagnostic Test: telephone interview — questionnaire PDEQ et IES-R

SUMMARY:
In France The prevalence of Pregnancy Loss after 12 weeks of gestation is around 3%. This situation is probably associated to a risk of post-traumatic stress disorder.

As a part of the medical staff midwives are often confronted with this situation, however they can have difficulties to identify short and long term effects of a post-traumatic stress disorders.

The purpose of the present study is to estimate and analyze the prevalence of short-term (1 month) post-traumatic stress disorder in women with pregnancy loss after 12 weeks of gestation.The symptoms of post-traumatic stress disorder will be tracked using the Impact of Event Scale-revisited and the Peritraumatic Dissociative Experiences Questionnaires.The diagnosis of post-traumatic stress disorder will also be clinically confirmed by a psychiatrist during a specific consultation.

ELIGIBILITY:
Inclusion Criteria:

* loss pregnancy after 12 weeks of gestation
* consent to participate in the clinical study

Exclusion Criteria:

* no french speaking
* psychiatric disease
* participation in another clinical study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Assessment of short-term post-traumatic stress disorder in women with fetal loss after 12 weeks of gestation with IES-R scale recorded at 30 days after fetal loss. | Telephone interviews are planned 30 days after fetal loss
  Assessment of the Impact of Events Scale-Revised (IES-R) score wil be performed by telephone interview by the principal investigator of the present study.
  IES-R scale has been validated in 1997 (Weiss and Mar) and then validated in French in 2003 (Brunet and St Hilaire). This scale assesses the semi-retarded and retarded consequences of traumatic events. It consists in a 22 items questionnaire measuring symptoms of post-traumatic stress disorder (PTSD), just after traumatic event and after a while. It is based on three main PTSD's elements: avoidance symptoms (items 8, 11, 12, 13, 17, 22), intrusion symptoms (items 1, 3, 5, 6, 9, 16) and hyperarousal (items 2, 4, 10, 14, 15, 18, 21).The patient has to respond using Likert's scale.
  score interpretations: 24-32: those with scores this high who do not have full PTSD will have partial PTSD. >33 this represents the best cutoff for a probable diagnosis of PTSD

CONTACTS AND LOCATIONS:
Overall Officials: lucile Abiola, Principal Investigator — Principal Investigator
Locations (1):
- CHU Angers, Angers, France

REFERENCES:
- [Derived] Abiola L, Legendre G, Spiers A, Parot-Schinkel E, Hamel JF, Duverger P, Bouet PE, Descamps P, Quelen C, Gillard P, Riquin E. Late fetal demise, a risk factor for post-traumatic stress disorder. Sci Rep. 2022 Jul 20;12(1):12364. doi: 10.1038/s41598-022-16683-5. PMID 35859001